CLINICAL TRIAL: NCT00402090
Title: Prevention of Thiopurines Related Toxicity Through the Determination by DHPLC TPMT Polymorphisms in Patients With ALL.
Brief Title: DHPLC Determination of TPMT Polymorphisms.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Cancerología (Other Government)
Other Study IDs: 005/007/ICI; CONACYT: Salud-2004-01-005
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2006-11-22 (Estimated); Status verified 2006-11

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: thiopurines; thiopurine methyl transferase; toxicity; pharmacogenomics
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
TPMT is a key enzyme in the metabolism of thiopurines. TPMT polymorphisms have been described and are associated with a decrease activity of such enzyme. Therefore, a higher risk of developing toxicity is present in patients requiring these drugs, which are indicated in acute lymphoblastic leukemia, as well as, immunosuppressors after organ transplantation. The frequency of heterozygotes polymorphisms ranges from 3 till 12 %, in different populations. Homozygous patients have a lower frequency, estimated 1 in 300 individuals. The frequency of such polymorphisms in mestizos mexican population has not been analyzed, and we considered important to determine this frequency in healthy and patients requiring thiopurines, particularly acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
Objectives: Determine by DHPLC analysis the frequency of TPMT polymorphisms in mestizos mexican population with acute lymphoblastic leukemia.

* To do a clinical correlation between the presence of polymorphism and thiopurine related- myelotoxicity.
* Inclusion criteria: Healthy volunteers or patients with acute lymphoblastic leukemia, age > 18 years, who attend to the National Institute of Cancerologia.
* Exclussion criteria: Patients with ALL, who are unable to have an adequate follow-up.
* Samples: Genomic DNA from peripheral blood leukocytes was isolated by standard methods. Known (wild-type and polymorphic) sequenced polymerase chain reaction (PCR) fragments of the TPMT gene were used as controls. TPMT gene fragments were amplified. PCR products were then analyzed by denaturating high performance liquid chromatography (DHPLC).

ELIGIBILITY:
Inclusion Criteria:

* Healthy and patientes with acute lymphoblastic leukemia.
* Age: older than 18 years.
* Attend to the National Institute of Cancerologia

Exclusion Criteria:

* Foreign patients with an irregular attendance to the National Institute of Cancerologia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-04; Study Completion 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Myrna Candelaria, MD, Principal Investigator — National Institute of Cancerologia
Locations (1):
- National Institute of Cancerologia, Mexico City, Mexico City, Mexico